CLINICAL TRIAL: NCT00419731
Title: Phase II Randomized, Double-Blind Trial of Bupropion Versus Bupropion + Naltrexone for Smoking Cessation
Brief Title: Study of Bupropion Versus Bupropion + Naltrexone for Smoking Cessation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Marc E. Mooney, Ph.D., University of Minnesota
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K01DA019446-01 (NIH); K01DA019446-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine; smoking; addiction
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Behavior, Addictive | interventions — Bupropion; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bupropion+Placebo
  Interventions: Drug: Bupropion
- 2 (Experimental): Bupropion+Naltrexone
  Interventions: Drug: Bupropion + Naltrexone

INTERVENTIONS:
Drug: Bupropion — Sustained-release, 150 mg, q.d., for days 1-3, 150 mg, b.i.d., for balance of 7 weeks.
  Placebo, 25 mg, q.d., for 7 weeks.
  Arms: 1
Drug: Bupropion + Naltrexone — Bupropion, Sustained-release, 150 mg, q.d., for days 1-3, 150 mg, b.i.d., for balance of 7 weeks.
  Naltrexone, 25 mg, q.d., for 7 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of bupropion + placebo to bupropion + naltrexone as treatments to help smokers quit.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of bupropion + placebo to bupropion + naltrexone as treatments to help smokers quit. Bupropion is an FDA-approved medication for smoking cessation that is believed to provide relief from craving and withdrawal through promotion of two neurotransmitter chemicals, dopamine and noradrenaline. Naltrexone is an FDA-approved medication for the treatment of opiate and alcohol dependence, that appears to function through blocking certain opiate receptors in the brain. It is expected that bupropion + naltrexone will produce higher smoking quit rates than bupropion + placebo. Bupropion alone is effective in alleviating some nicotine withdrawal complaints and craving for nicotine. However, bupropion does not reduce the rewarding effects of slips to smoking. Naltrexone alone is not generally effective as a smoking cessation medication, but it does help to reduce the rewarding effects of slips to smoking. Thus, it may help to prevent full relapse to smoking. In addition, naltrexone can help to reduce craving for cigarettes. It is hypothesized that the differing complementary actions of the two drugs will help smokers more than bupropion alone. In addition to examining smoking quit rates, the proposed study will also look at psychological processes that change during smoking cessation including, nicotine withdrawal, nicotine craving, mood, impulsivity, and attention

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Smoked at least 10 cigarettes/day for at least 1 year.
* English speaking.
* Females who are of childbearing potential must practice effective contraception and meet the following criteria:
* Are instructed to avoid pregnancy through 30 days after the last dose of study medication.
* Have a negative urine pregnancy test at baseline.
* Agree to use of the birth control methods listed: an oral contraceptive agent, an intrauterine device (IUD), an implantable contraceptive (e.g., Norplant), or an injectable contraceptive (e.g., Depo-Provera) for at least one month prior to entering the study and will continue its use through at least 30 days after the last dose of the study medication. A barrier method of contraception (e.g., condom or diaphragm with spermicide) while participating in the study and 30 days after the last dose of study medication.
* Willingness to reduce alcohol consumption during study to 2 or fewer standard drinks/day (3 oz. of alcohol or two beers (12 oz.), or two 5 oz. glasses of wine).
* Willingness to not use illicit drugs during study period including marijuana.

Exclusion Criteria:

* Concurrent use of tobacco products (other than cigarettes) or nicotine products.
* Contraindications to use of bupropion (i.e., concurrent use of other forms of bupropion, MAO inhibitors, anti-depressant medication, seizure disorder or any clinical situation that might increase risk for seizures, past head injury, current or prior diagnosis of bulimia or anorexia nervosa; bipolar disorder).
* Contraindications to use of naltrexone (i.e., past history of opioid abuse or dependence or evidence of opioid use in the past 30 days; significant hepatocellular injury as evidenced by liver enzyme levels over 3 times normal limits).
* Use of medications whose metabolism or effects may be adversely altered by bupropion or naltrexone. Medications that contraindicate the use of bupropion include theophylline, procarbazine, carbimazole, nialamide, pargyline, toloxatone, iproniazid, and systemic steroids. Medications that contraindicate the use of naltrexone include opioid analgesics and yohimbine.
* Current use of anti-seizure medications, disulfiram, or any medications that significantly challenge liver functioning.
* Treatment for drug or alcohol dependence during the last year, or evidence of alcohol abuse so severe that the patient is judged potentially unable to comply with the protocol.
* Evidence of problem alcohol consumption based on AUDIT.
* Self-reported use of illicit drugs in the past 90 days (including opioids, but excluding marijuana).
* Suicidal or homicidal ideation.
* Current major depression.
* History of bipolar disorder.
* Recent (within twelve months) myocardial infarction.
* Pregnant or lactating or planning pregnancy during treatment period.
* Having plans to leave the immediate geographical area within 9 months.
* Unwillingness or inability to given written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-02 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Biochemically-verified point-prevalence abstinence | 7, 11, 16, and 30 weeks post-quit
Likelihood of progression to a relapse (e.g., return to baseline smoking) following a slip at any time in study. | At any point following the quit date.
Treatment completion. | Weeks 7 and 30.
Daily cigarette smoking rate. | Weekly
Frequency and severity of bupropion and naltrexone side effects. | Weekly during treatment

SECONDARY OUTCOMES:
Attentional bias. | Weeks 1, 3, and 7.
Impulsivity. | Weeks 1, 3, and 7.
Nicotine withdrawal, craving and negative/positive affect. | All visits.

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Mooney, Ph.D., Principal Investigator — Univerisity of Minnesota
Locations (1):
- Tobacco Use Research Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Ascher JA, Cole JO, Colin JN, Feighner JP, Ferris RM, Fibiger HC, Golden RN, Martin P, Potter WZ, Richelson E, et al. Bupropion: a review of its mechanism of antidepressant activity. J Clin Psychiatry. 1995 Sep;56(9):395-401. PMID 7665537
- [Background] Mooney ME, Sofuoglu M. Bupropion for the treatment of nicotine withdrawal and craving. Expert Rev Neurother. 2006 Jul;6(7):965-81. doi: 10.1586/14737175.6.7.965. PMID 16831112
- [Background] Lerman C, Roth D, Kaufmann V, Audrain J, Hawk L, Liu A, Niaura R, Epstein L. Mediating mechanisms for the impact of bupropion in smoking cessation treatment. Drug Alcohol Depend. 2002 Jul 1;67(2):219-23. doi: 10.1016/s0376-8716(02)00067-4. PMID 12095672
- [Background] Shiffman S, Johnston JA, Khayrallah M, Elash CA, Gwaltney CJ, Paty JA, Gnys M, Evoniuk G, DeVeaugh-Geiss J. The effect of bupropion on nicotine craving and withdrawal. Psychopharmacology (Berl). 2000 Jan;148(1):33-40. doi: 10.1007/s002130050022. PMID 10663415
- [Background] Hutchison KE, Monti PM, Rohsenow DJ, Swift RM, Colby SM, Gnys M, Niaura RS, Sirota AD. Effects of naltrexone with nicotine replacement on smoking cue reactivity: preliminary results. Psychopharmacology (Berl). 1999 Feb;142(2):139-43. doi: 10.1007/s002130050872. PMID 10102765
- [Background] Wong GY, Wolter TD, Croghan GA, Croghan IT, Offord KP, Hurt RD. A randomized trial of naltrexone for smoking cessation. Addiction. 1999 Aug;94(8):1227-37. doi: 10.1046/j.1360-0443.1999.948122713.x. PMID 10615738
- [Background] Krishnan-Sarin S, Meandzija B, O'Malley S. Naltrexone and nicotine patch smoking cessation: a preliminary study. Nicotine Tob Res. 2003 Dec;5(6):851-7. doi: 10.1080/14622200310001614601. PMID 14750508
- [Background] Williams J, Ziedonis DM. Naltrexone-bupropion combination therapy for protracted abstinence dysphoria. Am J Addict. 2003 May-Jun;12(3):270-2. No abstract available. PMID 12851023
- [Background] Epstein AM, King AC. Naltrexone attenuates acute cigarette smoking behavior. Pharmacol Biochem Behav. 2004 Jan;77(1):29-37. doi: 10.1016/j.pbb.2003.09.017. PMID 14724039
- [Background] King A, de Wit H, Riley RC, Cao D, Niaura R, Hatsukami D. Efficacy of naltrexone in smoking cessation: a preliminary study and an examination of sex differences. Nicotine Tob Res. 2006 Oct;8(5):671-82. doi: 10.1080/14622200600789767. PMID 17008194
- [Background] King AC, Meyer PJ. Naltrexone alteration of acute smoking response in nicotine-dependent subjects. Pharmacol Biochem Behav. 2000 Jul;66(3):563-72. doi: 10.1016/s0091-3057(00)00258-6. PMID 10899371
- [Background] Brauer LH, Behm FM, Westman EC, Patel P, Rose JE. Naltrexone blockade of nicotine effects in cigarette smokers. Psychopharmacology (Berl). 1999 Apr;143(4):339-46. doi: 10.1007/s002130050957. PMID 10367550
- [Background] Ahmadi J, Ashkani H, Ahmadi M, Ahmadi N. Twenty-four week maintenance treatment of cigarette smoking with nicotine gum, clonidine and naltrexone. J Subst Abuse Treat. 2003 Apr;24(3):251-5. doi: 10.1016/s0740-5472(03)00027-8. PMID 12810146
- [Background] Sutherland G, Stapleton JA, Russell MA, Feyerabend C. Naltrexone, smoking behaviour and cigarette withdrawal. Psychopharmacology (Berl). 1995 Aug;120(4):418-25. doi: 10.1007/BF02245813. PMID 8539322
- [Background] Wewers ME, Dhatt R, Tejwani GA. Naltrexone administration affects ad libitum smoking behavior. Psychopharmacology (Berl). 1998 Nov;140(2):185-90. doi: 10.1007/s002130050756. PMID 9860109
- [Background] Covey LS, Glassman AH, Stetner F. Naltrexone effects on short-term and long-term smoking cessation. J Addict Dis. 1999;18(1):31-40. doi: 10.1300/J069v18n01_04. PMID 10234561
- [Background] Lerner AG, Oyffe I, Sigal M. Naltrexone-induced reduction of tobacco intake. J Clin Psychiatry. 1998 Jan;59(1):30-1. doi: 10.4088/jcp.v59n0107c. No abstract available. PMID 9491065
- [Background] David S, Lancaster T, Stead LF. Opioid antagonists for smoking cessation. Cochrane Database Syst Rev. 2001;(3):CD003086. doi: 10.1002/14651858.CD003086. PMID 11687036
- [Background] Toll BA, Leary V, Wu R, Salovey P, Meandzija B, O'Malley SS. A preliminary investigation of naltrexone augmentation of bupropion to stop smoking with less weight gain. Addict Behav. 2008 Jan;33(1):173-9. doi: 10.1016/j.addbeh.2007.05.012. Epub 2007 Jun 2. PMID 17587504
- [Background] Plodkowski RA, Nguyen Q, Sundaram U, Nguyen L, Chau DL, St Jeor S. Bupropion and naltrexone: a review of their use individually and in combination for the treatment of obesity. Expert Opin Pharmacother. 2009 Apr;10(6):1069-81. doi: 10.1517/14656560902775750. PMID 19364254
- [Derived] Mooney ME, Schmitz JM, Allen S, Grabowski J, Pentel P, Oliver A, Hatsukami DK. Bupropion and naltrexone for smoking cessation: A double-blind randomized placebo-controlled clinical trial. Clin Pharmacol Ther. 2016 Oct;100(4):344-52. doi: 10.1002/cpt.402. Epub 2016 Jun 20. PMID 27213949